CLINICAL TRIAL: NCT03810963
Title: Electrically Induced Cycling and Nutritional Counseling for Counteracting Obesity After SCI
Brief Title: FES Cycling and Nutritional Counseling for Battling Obesity After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Carey University (Other)
Collaborators: University of Southern Mississippi (Other); University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, David Dolbow, Associate Professor of Physical Therapy, William Carey University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WilliamCareyU
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injuries
Keywords: High intensity interval training; functional electrical stimulation cycling; chronic spinal cord injury; cardiometabolic disease risk; body composition; body fat percentage; nutritional counseling
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: The hypothesis for our research aim is that combining RG-HIIT-FES cycling with nutritional counseling will be more effective than nutritional counseling alone for reducing obesity and enhancing cardiometabolic health markers in persons with chronic SCI. This will be tested using a subject-matched controlled pre-post design. The experimental group receives 30 minutes of RG-HIIT-FES cycling three times per week for eight weeks and nutritional counseling over the telephone for 30 minutes one time per week for eight weeks. The control group receives the nutritional counseling only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES Cycling and Nutrition Counseling (Experimental): Device:
  HIIT-FES cycling will be performed 30 minutes per session, 3 times per week for 3 weeks combined with
  Behavior:
  Nutrition counseling will be completed via telephone for 30 minutes once per week for 8 weeks.
  Interventions: Combination Product: HIIT-FES Cycling combined with Nutritional Counseling
- Nutritional Counseling Only (Other): Behavior:
  Nutritional counseling will be completed via telephone for 30 minutes once per week for 8 weeks.
  Interventions: Other: Nutritional Counseling Only

INTERVENTIONS:
Combination Product: HIIT-FES Cycling combined with Nutritional Counseling — High intensity interval training functional electrical stimulation cycling for 30 minutes, three days per week for eight weeks, Nutritional counseling over the telephone for 30 minutes once per week for eight weeks.
  Arms: FES Cycling and Nutrition Counseling
Other: Nutritional Counseling Only — Nutritional counseling over the telephone for 30 minutes once per week for eight weeks.
  Arms: Nutritional Counseling Only

SUMMARY:
Individuals who suffer from paralysis after spinal cord injury (SCI) are estimated to have an even greater (66%) prevalence of obesity. Obesity is a major public health concern and is associated with a plethora of cardiometabolic health complications (heart disease, stroke and type II diabetes mellitus). Although the benefits of physical activity to counteract obesity and cardiometabolic disease have been documented, SCI typically limits voluntary exercise to the often injured arms (60-90%). On the other hand, functional electrical stimulation (FES) cycling has proven to be a safe and effective way to exercise paralyzed leg muscles in clinical and home settings, saving the often overworked arms. The investigators have developed a novel high-intensity interval training (HIIT) protocol for FES lower extremities cycling that may provide equal or greater benefits with less time commitment. The investigators proof-of-principle study in 3 obese persons with SCI confirmed that HIIT-FES cycling 3 times per week for 8 weeks without dietary monitoring can increase legs lean mass (5-9%), increase cardiovascular health markers (58% on average) and decrease HbA1c blood levels (2-4%). Also, 2 persons decreased body weight and BMI. The investigators hypothesize that combining HIIT-FES cycling with nutritional counseling will be effective for reducing obesity and enhancing cardiometabolic health in persons with chronic SCI. Research AIM: To determine preliminary efficacy of HIIT-FES cycling combined with nutritional counseling in obese adults with SCI. In this pilot two-arm, parallel, pre-post, subject-matched controlled trial, we will test the hypothesis that the experimental group receiving HIIT-FES cycling plus nutritional counseling will decrease total body weight, decrease body fat percentage, decrease fat mass, increase total and legs lean mass, improve blood lipid levels, decrease blood glucose and HbA1c levels and improve vascular endothelial health (flow mediated dilation) significantly more than age-, sex- and injury-matched controls receiving nutritional counseling only. The investigators will recruit 20 obese adults, 21-65 years of age, with chronic post-traumatic SCI ranging in neurological level between C4 and T12. Participants will be divided into experimental (HIIT-FES cycling plus nutritional counseling) and control (nutritional counseling only) groups.

DETAILED DESCRIPTION:
Obesity prevalence among individuals with SCI is about 66%. However, when the BMI formula is adjusted for the loss of muscle after SCI, the combined overweight and obesity rate is 70 to 75%. This places the SCI population across the U.S. at the top of the list in terms of obesity. Additionally, because greater obesity is related to greater disability and chronic diseases, the risk of cardiometabolic diseases, including heart disease, stroke and type II diabetes, are elevated to more than twice that of the able-bodied population. One reason for high obesity after SCI is the loss of muscle mass. Shortly after injury, those with SCI experience rapid and significant skeletal muscle atrophy below the level of injury resulting in skeletal muscle cross-sectional areas of 45-80% less than that of able-bodied individuals. Therefore, after SCI, the loss of metabolically active muscle mass results in a 26% reduction in basal metabolic rate and resting energy expenditure. This is important because basal metabolic rate accounts for ~65% of the total daily energy expenditure after SCI. In addition to decreased muscle mass, individuals with SCI are typically among the most sedentary, thus further lowering energy expenditure creating an unhealthy energy balance.

The benefits of physical activity for reducing obesity and cardiometabolic disease have been well documented. In particular, high-intensity interval training (HIIT) has been shown to decrease cardiovascular and metabolic risk among able-bodied individuals in a shorter period of time than standard non-interval exercise programs. For example, one comparison of interval walking to continuous walking in able-bodied adults with type II diabetes over a 6-month period. The continuous walking group walked for 60 minutes 5 days per week at a moderate intensity while the interval training group alternated between 3 minutes of high intensity walking and 3 minutes of low intensity walking 5 days per week. The walking intensities were determined by oxygen uptake (VO2) peak testing and energy expenditure, with moderate intensity being set at 55% and high intensity at 70% of VO2 peak. Although, the mileage was the same for both groups, the interval training group lost 4.3 ± 1.2 kg total body weight and 3.1 ± 0.7 kg body fat mass, whereas no changes in body composition were found in the continuous walking group or the non-walking control group. In a similar study, another researcher used leg cycling 3 times per week for 12 weeks in both the continuous and interval groups and determined intensity levels based on heart rate. The interval training group performed 3 "all out" cycling sessions of 20 seconds each separated by 2 minutes low intensity cycling, while the continuous group cycled steady at 70% of maximal heart rate for 45 minutes. Both groups improved similarly in insulin sensitivity, cardiorespiratory fitness, and skeletal muscle mitochondrial content, however, the interval training group achieved these benefits with a five-fold lower exercise volume and training time commitment.

A major consequence of SCI is that paralysis makes voluntary exercise with the legs impossible. In addition, the 60-90% prevalence of shoulder pain in persons with chronic SCI is often limiting the possibility of regular arm exercise. To circumvent these problems, FES has been shown to be a safe and effective way to exercise paralyzed leg muscles in clinical and home settings. High-cadence moderate-resistance FES cycling can increase muscle mass and improve fasting blood glucose values and low-cadence higher-resistance FES cycling can lead to hypertrophy of the paralyzed leg muscles. As a result of developing our new protocol, which incorporates resistance-guided high-intensity interval training into FES cycling (RG-HIIT-FES), we postulate that it may provide equal or greater benefits with less exercise time commitment, by analogy to high-intensity interval training programs used by able-bodied individuals. The advantage of using resistance as the determinant of exercise intensity is the fact that heart rate is an ineffective method for monitoring exercise intensity after SCI. Instead, we first determine the greatest resistance that stimulated muscles can work against while cycling at 35 rpm for 30 seconds, use 80% of that maximal resistance for the high-intensity cycling interval (30 seconds), and then decrease it to 0.5 Nm, which is the lowest resistance provided by the FES bike (RT300) for the low-intensity cycling interval (30 seconds). These intervals are then alternated for 30 minutes. In a proof-of-principle case series study using this RG-HIIT-FES cycling protocol 3 times per week for 8 weeks, 3 obese individuals with SCI increased legs lean mass (5-9%), improved vascular endothelial health (mean increase of 58% in arterial flow mediated dilation), and decreased HbA1c blood levels (2-4%). Two of the three participants decreased body weight and BMI.

It is important for proper interpretation of results not to overlook the significance of nutritional counseling concerning energy intake because food intake can have a major effect on body composition and health. Individuals with SCI are especially in need of nutritional counseling due to decreased energy expenditure from reduced metabolic muscle and decreased activity levels. Consequently, our central hypothesis is that a combined program of RG-HIIT-FES cycling and nutritional counseling will be effective in combating obesity and enhancing cardiometabolic health for those with SCI. Specifically, decrease total body weight and percent body fat, increase total and legs lean mass, improve blood lipid levels, decrease blood glucose and HbA1c levels and improve cardiovascular health markers (arterial flow mediated dilation) beyond that observed in the control group that will receive nutritional counseling alone. The intervention group will receive three 30-minute RG-HIIT-FES cycling sessions and one 30-minute nutritional counseling session per week for 8 weeks, whereas the control group will receive one 30-minute nutritional counseling session per week for 8 weeks.

Innovation: The proposed pilot study provides at least three important innovations: 1) the first formal implementation of a novel and promising FES cycling protocol (RG-HIIT-FES); 2) the first testing of potential benefits of combining FES cycling with nutritional counseling in any population; 3) enrollment of a medically underserved and disadvantaged population with limited options for battling obesity and maintaining cardiovascular health.

Planned Experimental Protocols: The hypothesis for our research aim is that combining RG-HIIT-FES cycling with nutritional counseling will be more effective than nutritional counseling alone for reducing obesity and enhancing cardiometabolic health markers in persons with chronic SCI. This will be tested using a subject-matched controlled pre-post design. Prior to and after the 8 weeks of experimental or control intervention, each participant will visit the SCI Research Laboratory during the morning hours (between 7:00 and 10:00 am), following an overnight fast and having refrained from caffeine and alcohol intake for 12 and 24 hours, respectively. After reviewing and signing the informed consent and medical history documents, participants will be weighed using a Scale-Tronix Wheelchair Scale (Welch Allyn, Skaneatelest Falls, NY). The weight of the wheelchair alone subtracted from the combined weight of the participant and wheelchair will provide the weight of the participant. An electric powered lift (Invacare, Reliant 450) will be used to provide safe transfers for all participants from the participant's wheelchair to various testing locations (e.g., exam table and DXA body composition scanner). Once on the exam table in a supine position, an anthropometric measuring rod will be used to measure height. The left leg will be extended and ankle dorsiflexed to enable an accurate measurement from the bottom of foot to top of the head. Following 20 minutes of quiet rest in a dimly lit and temperature (21-23°C, 50% humidity) controlled room, 5 minutes of resting hemodynamic data (hear rate and blood pressure) will be recorded followed by Doppler ultrasound vascular endothelial function testing, followed shortly after by a finger stick on the left hand for determination of blood lipid, glucose and HbA1c levels. The participants will then be transferred back to their wheelchair and taken to an adjacent laboratory in the same building for DXA scanning. Following the DXA scan, participants return to the SCI Research lab and complete a resistance guided FES cycle maximal test from there own wheelchairs in order to gain baseline parameters for the RG-HIIT-FES cycling protocol, and also to determine each participants ability to tolerate and safely perform the cycling program. Participants in the experimental/intervention group will then complete FES cycling as described above for 30 minutes, 3 times per week for 8 weeks and will receive nutritional counseling over the telephone for 30 minutes 1 time per week for 8 weeks. Then post-testing will occur in the same fashion as the pre-testing.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit men and women with C4-T12 SCI (n=20) American Spinal Injury Association Impairment Scale A, B, or C as per International Standards for Neurological Classification of SCI; ≥2 years post-SCI; age 21-65 years; body fat percentage according to over-weight classifications detailed in Gallagher et al. Am J Clin Nut 2000,72:694-701 ( women 20-40 y/o > 30%, 41-60 y/o > 35%, > 60 y/o > 42%; men 20-40 y/o > 19%, 40-60 y/o > 22%, > 60 y/o > 25%).

Exclusion Criteria:

* Exclusion criteria include pressure wounds on buttocks or feet; unhealed bone fractures or history of fragility fractures; uncontrolled cardiovascular or metabolic disease; severe osteoporosis (T score ≤ 4); uncontrolled autonomic dysreflexia; and current smokers.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage | Eight Weeks
  Percentage of body fat measured during pre- and post-testing
Fat mass and lean mass | Eight Weeks
  Total fat and lean mass in kg measured during pre- and post-testing
Arterial health via flow mediated dilation | Eight Weeks
  Measurement of arterial diameter change in mm after blood flow restriction during pre- poste testing
Blood glucose testing | 8 weeks
  Using finger stick blood droplet method pre- and post-testing for blood glucose and HbA1c measures

SECONDARY OUTCOMES:
Pre- post- intervention three day dietary recall | Eight Weeks
  Prior to and after the intervention a 3 day dietary recall will be completed to determine changes in dietary habits.

CONTACTS AND LOCATIONS:
Overall Officials: David Dolbow, DPT, PhD, Principal Investigator — William Carey University
Locations (1):
- William Carey University Physical Therapy Program, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
None currently

REFERENCES:
- [Background] Conway JM, Ingwersen LA, Moshfegh AJ. Accuracy of dietary recall using the USDA five-step multiple-pass method in men: an observational validation study. J Am Diet Assoc. 2004 Apr;104(4):595-603. doi: 10.1016/j.jada.2004.01.007. PMID 15054345
- [Result] Froehlich-Grobe K, Lee J, Washburn RA. Disparities in obesity and related conditions among Americans with disabilities. Am J Prev Med. 2013 Jul;45(1):83-90. doi: 10.1016/j.amepre.2013.02.021. PMID 23790992
- [Result] Gater DR Jr. Obesity after spinal cord injury. Phys Med Rehabil Clin N Am. 2007 May;18(2):333-51, vii. doi: 10.1016/j.pmr.2007.03.004. PMID 17543776
- [Result] Rajan S, McNeely MJ, Warms C, Goldstein B. Clinical assessment and management of obesity in individuals with spinal cord injury: a review. J Spinal Cord Med. 2008;31(4):361-72. doi: 10.1080/10790268.2008.11760738. PMID 18959353
- [Result] Laughton GE, Buchholz AC, Martin Ginis KA, Goy RE; SHAPE SCI Research Group. Lowering body mass index cutoffs better identifies obese persons with spinal cord injury. Spinal Cord. 2009 Oct;47(10):757-62. doi: 10.1038/sc.2009.33. Epub 2009 Apr 7. PMID 19350042
- [Result] Gorgey AS, Dolbow DR, Dolbow JD, Khalil RK, Gater DR. The effects of electrical stimulation on body composition and metabolic profile after spinal cord injury--Part II. J Spinal Cord Med. 2015 Jan;38(1):23-37. doi: 10.1179/2045772314Y.0000000244. Epub 2014 Jul 8. PMID 25001669
- [Result] Cragg JJ, Noonan VK, Krassioukov A, Borisoff J. Cardiovascular disease and spinal cord injury: results from a national population health survey. Neurology. 2013 Aug 20;81(8):723-8. doi: 10.1212/WNL.0b013e3182a1aa68. Epub 2013 Jul 24. PMID 23884034
- [Result] Groah SL, Nash MS, Ward EA, Libin A, Mendez AJ, Burns P, Elrod M, Hamm LF. Cardiometabolic risk in community-dwelling persons with chronic spinal cord injury. J Cardiopulm Rehabil Prev. 2011 Mar-Apr;31(2):73-80. doi: 10.1097/HCR.0b013e3181f68aba. PMID 21045711
- [Result] Eriks-Hoogland IE, Hoekstra T, de Groot S, Stucki G, Post MW, van der Woude LH. Trajectories of musculoskeletal shoulder pain after spinal cord injury: Identification and predictors. J Spinal Cord Med. 2014 May;37(3):288-98. doi: 10.1179/2045772313Y.0000000168. Epub 2013 Nov 7. PMID 24621031
- [Result] Alm M, Soroudi N, Wylie-Rosett J, Isasi CR, Suchday S, Rieder J, Khan U. A qualitative assessment of barriers and facilitators to achieving behavior goals among obese inner-city adolescents in a weight management program. Diabetes Educ. 2008 Mar-Apr;34(2):277-84. doi: 10.1177/0145721708314182. PMID 18375777
- [Result] Medina GI, Nascimento FB, Rimkus CM, Zoppi Filho A, Cliquet A Jr. Clinical and radiographic evaluation of the shoulder of spinal cord injured patients undergoing rehabilitation program. Spinal Cord. 2011 Oct;49(10):1055-61. doi: 10.1038/sc.2011.64. Epub 2011 Jul 5. PMID 21727901
- [Result] Jain NB, Higgins LD, Katz JN, Garshick E. Association of shoulder pain with the use of mobility devices in persons with chronic spinal cord injury. PM R. 2010 Oct;2(10):896-900. doi: 10.1016/j.pmrj.2010.05.004. PMID 20970758
- [Result] Brose SW, Boninger ML, Fullerton B, McCann T, Collinger JL, Impink BG, Dyson-Hudson TA. Shoulder ultrasound abnormalities, physical examination findings, and pain in manual wheelchair users with spinal cord injury. Arch Phys Med Rehabil. 2008 Nov;89(11):2086-93. doi: 10.1016/j.apmr.2008.05.015. PMID 18996236
- [Result] Curtis KA, Drysdale GA, Lanza RD, Kolber M, Vitolo RS, West R. Shoulder pain in wheelchair users with tetraplegia and paraplegia. Arch Phys Med Rehabil. 1999 Apr;80(4):453-7. doi: 10.1016/s0003-9993(99)90285-x. PMID 10206610
- [Result] Dolbow DR, Gorgey AS, Ketchum JM, Moore JR, Hackett LA, Gater DR. Exercise adherence during home-based functional electrical stimulation cycling by individuals with spinal cord injury. Am J Phys Med Rehabil. 2012 Nov;91(11):922-30. doi: 10.1097/PHM.0b013e318269d89f. PMID 23085704
- [Result] Griffin L, Decker MJ, Hwang JY, Wang B, Kitchen K, Ding Z, Ivy JL. Functional electrical stimulation cycling improves body composition, metabolic and neural factors in persons with spinal cord injury. J Electromyogr Kinesiol. 2009 Aug;19(4):614-22. doi: 10.1016/j.jelekin.2008.03.002. Epub 2008 Apr 25. PMID 18440241
- [Result] Fornusek C, Davis GM, Russold MF. Pilot study of the effect of low-cadence functional electrical stimulation cycling after spinal cord injury on thigh girth and strength. Arch Phys Med Rehabil. 2013 May;94(5):990-3. doi: 10.1016/j.apmr.2012.10.010. Epub 2012 Oct 30. PMID 23123504
- [Result] DeVivo MJ, Krause JS, Lammertse DP. Recent trends in mortality and causes of death among persons with spinal cord injury. Arch Phys Med Rehabil. 1999 Nov;80(11):1411-9. doi: 10.1016/s0003-9993(99)90252-6. PMID 10569435
- [Result] Labounty TM, Gomez MJ, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng V, Chinnaiyan KM, Chow B, Cury R, Delago A, Dunning A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann P, Kim YJ, Leipsic J, Lin FY, Maffei E, Raff G, Shaw LJ, Villines TC, Min JK. Body mass index and the prevalence, severity, and risk of coronary artery disease: an international multicentre study of 13,874 patients. Eur Heart J Cardiovasc Imaging. 2013 May;14(5):456-63. doi: 10.1093/ehjci/jes179. Epub 2012 Aug 24. PMID 22922955
- [Result] Ramaswamy P, Chikkabyrappa S, Donda K, Osmolovsky M, Rojas M, Rafii D. Relationship of ambulatory blood pressure and body mass index to left ventricular mass index in pediatric patients with casual hypertension. J Am Soc Hypertens. 2016 Feb;10(2):108-14. doi: 10.1016/j.jash.2015.11.009. Epub 2015 Nov 22. PMID 26725015
- [Result] Winter Y, Rohrmann S, Linseisen J, Lanczik O, Ringleb PA, Hebebrand J, Back T. Contribution of obesity and abdominal fat mass to risk of stroke and transient ischemic attacks. Stroke. 2008 Dec;39(12):3145-51. doi: 10.1161/STROKEAHA.108.523001. Epub 2008 Aug 14. PMID 18703800
- [Result] Spungen AM, Adkins RH, Stewart CA, Wang J, Pierson RN Jr, Waters RL, Bauman WA. Factors influencing body composition in persons with spinal cord injury: a cross-sectional study. J Appl Physiol (1985). 2003 Dec;95(6):2398-407. doi: 10.1152/japplphysiol.00729.2002. Epub 2003 Aug 8. PMID 12909613
- [Result] Castro MJ, Apple DF Jr, Hillegass EA, Dudley GA. Influence of complete spinal cord injury on skeletal muscle cross-sectional area within the first 6 months of injury. Eur J Appl Physiol Occup Physiol. 1999 Sep;80(4):373-8. doi: 10.1007/s004210050606. PMID 10483809
- [Result] Gorgey AS, Dudley GA. Skeletal muscle atrophy and increased intramuscular fat after incomplete spinal cord injury. Spinal Cord. 2007 Apr;45(4):304-9. doi: 10.1038/sj.sc.3101968. Epub 2006 Aug 29. PMID 16940987
- [Result] Biering-Sorensen B, Kristensen IB, Kjaer M, Biering-Sorensen F. Muscle after spinal cord injury. Muscle Nerve. 2009 Oct;40(4):499-519. doi: 10.1002/mus.21391. PMID 19705475
- [Result] Monroe MB, Tataranni PA, Pratley R, Manore MM, Skinner JS, Ravussin E. Lower daily energy expenditure as measured by a respiratory chamber in subjects with spinal cord injury compared with control subjects. Am J Clin Nutr. 1998 Dec;68(6):1223-7. doi: 10.1093/ajcn/68.6.1223. PMID 9846850
- [Result] Yilmaz B, Yasar E, Goktepe S, Alaca R, Yazicioglu K, Dal U, Mohur H. Basal metabolic rate and autonomic nervous system dysfunction in men with spinal cord injury. Obesity (Silver Spring). 2007 Nov;15(11):2683-7. doi: 10.1038/oby.2007.320. PMID 18070759
- [Result] Buchholz AC, Pencharz PB. Energy expenditure in chronic spinal cord injury. Curr Opin Clin Nutr Metab Care. 2004 Nov;7(6):635-9. doi: 10.1097/00075197-200411000-00008. PMID 15534431
- [Result] Karstoft K, Winding K, Knudsen SH, Nielsen JS, Thomsen C, Pedersen BK, Solomon TP. The effects of free-living interval-walking training on glycemic control, body composition, and physical fitness in type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2013 Feb;36(2):228-36. doi: 10.2337/dc12-0658. Epub 2012 Sep 21. PMID 23002086
- [Result] Gillen JB, Martin BJ, MacInnis MJ, Skelly LE, Tarnopolsky MA, Gibala MJ. Twelve Weeks of Sprint Interval Training Improves Indices of Cardiometabolic Health Similar to Traditional Endurance Training despite a Five-Fold Lower Exercise Volume and Time Commitment. PLoS One. 2016 Apr 26;11(4):e0154075. doi: 10.1371/journal.pone.0154075. eCollection 2016. PMID 27115137
- [Result] Gorgey AS, Harnish CR, Daniels JA, Dolbow DR, Keeley A, Moore J, Gater DR. A report of anticipated benefits of functional electrical stimulation after spinal cord injury. J Spinal Cord Med. 2012 Mar;35(2):107-12. doi: 10.1179/204577212X13309481546619. PMID 22525324
- [Result] Khalil RE, Gorgey AS, Janisko M, Dolbow DR, Moore JR, Gater DR. The role of nutrition in health status after spinal cord injury. Aging Dis. 2013 Feb;4(1):14-22. Epub 2012 Nov 30. PMID 23423356
- [Result] Valent LJ, Dallmeijer AJ, Houdijk H, Slootman J, Janssen TW, Hollander AP, van der Woude LH. The individual relationship between heart rate and oxygen uptake in people with a tetraplegia during exercise. Spinal Cord. 2007 Jan;45(1):104-11. doi: 10.1038/sj.sc.3101946. Epub 2006 Jun 27. PMID 16801936
- [Result] Dolbow DR, Gorgey AS, Dolbow JD, Gater DR. Seat pressure changes after eight weeks of functional electrical stimulation cycling: a pilot study. Top Spinal Cord Inj Rehabil. 2013 Summer;19(3):222-8. doi: 10.1310/sci1903-222. PMID 23960706
- [Result] Gorgey AS, Poarch HJ, Dolbow DD, Castillo T, Gater DR. Effect of adjusting pulse durations of functional electrical stimulation cycling on energy expenditure and fatigue after spinal cord injury. J Rehabil Res Dev. 2014;51(9):1455-68. doi: 10.1682/JRRD.2014.02.0054. PMID 25803753
- [Result] Shim JS, Oh K, Kim HC. Dietary assessment methods in epidemiologic studies. Epidemiol Health. 2014 Jul 22;36:e2014009. doi: 10.4178/epih/e2014009. eCollection 2014. PMID 25078382
- [Result] Conway JM, Ingwersen LA, Vinyard BT, Moshfegh AJ. Effectiveness of the US Department of Agriculture 5-step multiple-pass method in assessing food intake in obese and nonobese women. Am J Clin Nutr. 2003 May;77(5):1171-8. doi: 10.1093/ajcn/77.5.1171. PMID 12716668
- [Result] Stoner L, Sabatier M, VanhHiel L, Groves D, Ripley D, Palardy G, McCully K. Upper vs lower extremity arterial function after spinal cord injury. J Spinal Cord Med. 2006;29(2):138-46. doi: 10.1080/10790268.2006.11753867. PMID 16739557
- [Result] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Result] Credeur DP, Mariappan N, Francis J, Thomas D, Moraes D, Welsch MA. Vasoreactivity before and after handgrip training in chronic heart failure patients. Atherosclerosis. 2012 Nov;225(1):154-9. doi: 10.1016/j.atherosclerosis.2012.08.013. Epub 2012 Sep 16. PMID 23010159
- [Result] Stoner L, McCully KK. Peak and time-integrated shear rates independently predict flow-mediated dilation. J Clin Ultrasound. 2012 Jul-Aug;40(6):341-51. doi: 10.1002/jcu.21900. Epub 2012 Mar 11. PMID 22407951
- [Result] Restaino RM, Holwerda SW, Credeur DP, Fadel PJ, Padilla J. Impact of prolonged sitting on lower and upper limb micro- and macrovascular dilator function. Exp Physiol. 2015 Jul 1;100(7):829-38. doi: 10.1113/EP085238. Epub 2015 Jun 10. PMID 25929229